CLINICAL TRIAL: NCT01496144
Title: Manual Therapy Followed by Specific Active Exercises Versus a Placebo Followed by Specific Active Exercises on the Improvement of Functional Disability in Patients With Chronic Non Specific Low Back Pain: a Randomized Controlled Trial
Brief Title: Manual Therapy on the Improvement of Functional Disability in Patients With Chronic Non Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Pierre Balthazard, Bachelor of sciences in physical therapy, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNS13DPD3-109903; FNS13DPD3-109903 (Other Grant/Funding Number: Swiss National Fund DORE)
Record Dates: First submitted 2011-12-16; First posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Chronic non specific low back pain; Manual therapy; Active exercises; Pain; Disability
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual therapy and active exercises (Experimental): Spinal manipulation /mobilisation
  Interventions: Procedure: Manual therapy and active exercises
- Detuned ultrasound and active exercises (Placebo Comparator)
  Interventions: Procedure: Detuned ultrasound and active exercises

INTERVENTIONS:
Procedure: Manual therapy and active exercises — Spinal manipulation/mobilisation (5-10 minutes), consisting of passive accessory intervertebral movements, muscle-energy techniques and high velocity, low amplitude dynamic thrust.
  Active exercises (20 minutes), consisting of mobility, stretching, strengthening and motor control exercises
  Other Names: Spinal mobilisation; Manipulation
  Arms: Manual therapy and active exercises
Procedure: Detuned ultrasound and active exercises — Electrotherapy device inactivated and ineffective. Active exercises, consisting of mobility, stretching, strengthening and motor control exercises
  Other Names: Electrotherapy
  Arms: Detuned ultrasound and active exercises

SUMMARY:
Background: Models have tried to explain the driving mechanisms behind chronic non specific low back pain (CNSLBP) in order to propose better appropriate conservative treatment. Altered responses at spinal and/or supraspinal level may affect the perception of pain and degree of disability of CNSLBP patients. Recent clinical recommendations still propose active exercises (AE) for CNSLBP. However, acceptance of exercises by patients may be limited by pain-related manifestations. Current evidences suggest manual therapy (MT) induces a short-term analgesic effect through neurophysiological mechanisms at peripheral, spinal and cortical levels. The aim of this study was first, to assess whether MT has an instant analgesic effect, and second, to compare the long-lasting effect on functional disability of MT followed by AE to sham therapy (ST) followed by AE. Methods: Forty-two CNSLBP patients without co-morbidities, randomly distributed into 2 treatment groups, received either spinal manipulation/mobilization (first intervention) plus AE (MT group; n = 22), or detuned ultrasound (first intervention) plus AE (ST group; n = 20). Eight therapeutic sessions were delivered over 4 to 8 weeks. Instant analgesic effect was obtained by measuring pain intensity (Visual Analogue Scale) before and immediately after the first intervention of each therapeutic session. Pain intensity, disability (Oswestry Disability Index) and fear-avoidance beliefs (Fear-Avoidance Beliefs Questionnaire) were determined before treatment, after the 8th therapeutic session, and at 3- and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* suffering from non specific low back pain with or without symptoms in the lower extremity for a period between 12 and 26 weeks
* can maintain the usual medication

Exclusion Criteria:

* spinal fracture or surgery within the previous 6 months
* pregnancy
* neoplasia
* spinal infection
* spinal inflammatory arthritis
* low back pain of visceral origin
* severe sensitive and/or motor radicular deficit from nerve root origin of less than 6 months
* score of 3/5 or more on the Waddell Score
* on sick leaves from work for 6 months or more
* psychiatric disorders
* opioid medication
* patient unable to collaborate (linguistic barrier; cognitive impairments)
* radiologic abnormalities other than degenerative disease
* clinical neurogenic claudication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale - VAS-pain | During treatment, over a period of 4 to 8 weeks
  self-report of clinical pain intensity, consisting of a 10 cm horizontal line scale on which is added the statements "no pain" on the left and "maximum intensity of pain" on the right

SECONDARY OUTCOMES:
Fear-avoidance beliefs (Fear-Avoidance Beliefs Questionnaire - FABQ) | Before randomization and untill 6 months after the end of treatment
  measures level of fear and avoidance beliefs about work and physical activity in patients with low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Dériaz, MD, PhD, Study Director — Institut de Recherche en Réadaptation et Clinique Romande de Réadaptation SUVACare, Sion, Switzerland
Locations (1):
- Département de l'appareil locomoteur (DAL), Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Ferreira ML, Ferreira PH, Latimer J, Herbert RD, Hodges PW, Jennings MD, Maher CG, Refshauge KM. Comparison of general exercise, motor control exercise and spinal manipulative therapy for chronic low back pain: A randomized trial. Pain. 2007 Sep;131(1-2):31-7. doi: 10.1016/j.pain.2006.12.008. Epub 2007 Jan 23. PMID 17250965
- [Background] Aure OF, Nilsen JH, Vasseljen O. Manual therapy and exercise therapy in patients with chronic low back pain: a randomized, controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2003 Mar 15;28(6):525-31; discussion 531-2. doi: 10.1097/01.BRS.0000049921.04200.A6. PMID 12642755
- [Background] Hemmila HM, Keinanen-Kiukaanniemi SM, Levoska S, Puska P. Long-term effectiveness of bone-setting, light exercise therapy, and physiotherapy for prolonged back pain: a randomized controlled trial. J Manipulative Physiol Ther. 2002 Feb;25(2):99-104. doi: 10.1067/mmt.2002.122329. PMID 11896377
- [Background] Niemisto L, Lahtinen-Suopanki T, Rissanen P, Lindgren KA, Sarna S, Hurri H. A randomized trial of combined manipulation, stabilizing exercises, and physician consultation compared to physician consultation alone for chronic low back pain. Spine (Phila Pa 1976). 2003 Oct 1;28(19):2185-91. doi: 10.1097/01.BRS.0000085096.62603.61. PMID 14520029
- [Background] Assendelft WJ, Morton SC, Yu EI, Suttorp MJ, Shekelle PG. Spinal manipulative therapy for low back pain. A meta-analysis of effectiveness relative to other therapies. Ann Intern Med. 2003 Jun 3;138(11):871-81. doi: 10.7326/0003-4819-138-11-200306030-00008. PMID 12779297
- [Derived] Balthazard P, de Goumoens P, Rivier G, Demeulenaere P, Ballabeni P, Deriaz O. Manual therapy followed by specific active exercises versus a placebo followed by specific active exercises on the improvement of functional disability in patients with chronic non specific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Aug 28;13:162. doi: 10.1186/1471-2474-13-162. PMID 22925609